CLINICAL TRIAL: NCT02823535
Title: iWin: Navigating Your Path to Well-Being
Brief Title: Iwin: Individual Well-Being Navigator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Collaborators: IMS Health (Other)
Responsible Party: Principal Investigator, Kerry E. Evers, Co-President & CEO, Pro-Change Behavior Systems
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 271201500061C-0-0-1 (NIH)
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Other Drug Substance Abuse
Keywords: military; veteran; military spouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iwin: Individual Well-Being Navigator (Experimental): Iwin intervention during 6-month intervention period plus study assessments at baseline, 6, and 9 months.
  Interventions: Behavioral: Iwin: Individual Well-Being Navigator
- Control group (No Intervention): Study assessments at baseline, 6 months, and 9 months, plus two short surveys unrelated to the study behaviors at 4 and 5 months.

INTERVENTIONS:
Behavioral: Iwin: Individual Well-Being Navigator — Immediately following the baseline assessment, the Intervention Group will receive a secure link to download the IWin app. The app provides three types of integrated interventions: 1) stage-matched feedback on the participant's risk behaviors as determined via the assessments; 2) up to two in app messages a day determined by a series of algorithms that control the timing, content, and cadence of the messages; and 3) up to two prompts a week to complete stage-matched activities that foster behavior change (e.g., quizzes, calculators, guided visualizations, info-graphics, testimonials, and more).
  Arms: Iwin: Individual Well-Being Navigator

SUMMARY:
The overarching objective of this proposal is to conduct a randomized trial to evaluate the effectiveness of the Individual Well-Being Navigator (Iwin) mobile application, a substance abuse prevention and well-being enhancement program designed specifically for military personnel, veterans, and military spouses. Iwin provides an innovative, tailored mobile application using best practices in behavior change science and innovative technology to assist users in preventing substance abuse and enhancing well-being by providing them with the most appropriate intervention content at the right time. It integrates Transtheoretical Model of Behavior Change based tailoring, in app messaging, stage of change matched activities, and engaging game-like features in a cutting edge multiple behavior change program. The efficacy of the Iwin program will be determined by tests of statistical significance indicating that participants in the Treatment condition had lower scores on an index of substance use and other behavioral risks. The overall design is a 2 group (treatment and control group) by 3 Occasions with repeated measures across occasions.

DETAILED DESCRIPTION:
The overarching objective of this project is to conduct a randomized trial to evaluate the effectiveness of the Individual Well-Being Navigator (Iwin) mobile application, a substance abuse prevention and well-being enhancement program designed specifically for military personnel, veterans, and military spouses.

Military personnel, veterans, and military spouses recruited will be asked to complete a series of screening questions on their personal mobile devices. An estimated 476 Personnel will need to be screened to arrive at an eligible sample of 238. Randomization of the eligible sample will occur within the online baseline assessment at the individual level as soon as a participant completes the Informed Consent form. Those randomized to the Control Group (n=119) will complete assessments at baseline, 6 months, and 9 months. Additionally, the control group will complete a short survey unrelated to the study behaviors at 4 and 5 months to match incentives given to the intervention group. Those randomized to the Intervention Group (n=119) will complete the same schedule of assessments as the control group and in addition will have access to the Iwin application (app) in between the baseline and 6 month assessments. The assessments include a variety of questions on health, wellness, substance use and well-being.

Users randomized into the intervention group will be able to download the Iwin app for free onto their personal device. The Pro-Change Iwin application has been built using the IMS Health AppNucleus™ Platform. AppNucleus is a patented, federally certified (FIPS 140-2, DIACAP MAC II Sensitive), secure application platform that enables Pro-Change to rapidly deploy secure mHealth solutions to users via web portal and commercial mobile technologies (such as iOS, Android, Windows Phone, Blackberry). The application provides an innovative, tailored program using best practices in behavior change science and innovative technology to assist users in preventing substance abuse and enhancing well-being by providing them with the most appropriate intervention content at the right time for their individual needs. It delivers assessments and tailored feedback immediately on eleven different risk behaviors as well as mobile interactive staged matched activities, engaging game-like features and in-app notifications on each behavior they are at risk for over the course of 6 months. The app will provide reminders for users to return to the program as set time points. Both intervention and control participants will receive e-mail reminders to complete follow-up assessments at 6 and 9 months.

PRIVACY

All information shared with us will be kept confidential to the extent provided by law. Names will not be connected to survey answers. Instead, a code will be used in place of a name in the research study records. Access to the research records will be limited to the research study team. The research records will be deleted three years after the submission of the final financial report in accordance with OMB Circular A-110.

To help us protect participant privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify a participant in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify a partcipant. There is one exception to the promise of confidentiality: if we see or are told that someone is planning to harm themselves or someone else, we will disclose this information to the proper authorities.

The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). A Certificate of Confidentiality does not prevent a participant or a member of their family from voluntarily releasing information about the participant or their involvement in this research. If an insurer, medical care provider, or other person obtains a participants written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Between 18 and 54 years of age
3. Member of the U.S. Military (active duty, active reservist), Veteran, Military Spouse (only one member of each household is eligible)
4. Have access to a mobile device with Internet connectivity
5. Comfortable using applications on a mobile device
6. Have access to an email account they check at least weekly.

Exclusion Criteria:

1. Pregnant
2. Significant head injury or other condition that could prevent using mobile device
3. Admitted to an inpatient mental health facility in the past two years
4. Suicidal ideation
5. Moderately severe depression - i.e., score of > 15 on the Patient Health Questionnaire-8 (PHQ-8)
6. Severe PTSD symptoms (PCL-5 score > 61).

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Health Risk Behaviors Index | Baseline, 6 and 9 months
  Assesses risk status and stage of change for eleven health risk behaviors including: smoking, alcohol (risky drinking), financial well-being, other substance use, stress management, pain management, depression management, sleep management, regular exercise). Previous research has used this measure as an indicator of the effectiveness of an intervention for overall multiple behavior change.

SECONDARY OUTCOMES:
The Assist | Baseline, 6 and 9 months
  The ASSIST (Alcohol, Smoking, and Substance Involvement Screening Test) is an 8 item questionnaire that takes about 5-10 minutes to complete. Originally developed by the World Health Organization primarily for use in primary care settings to identify patients who substance use may be classified as moderate level, it has been adapted in a range of studies for use in other populations and research . This tool has also been adapted by NIDA and published online as a tool for clinicians. It screens for problem or risky use of tobacco, alcohol, cannabis, cocaine, ATS, sedatives, hallucinogens, inhalants, opioids, and other drugs. A risk score is developed for each category, as well as an overall risk score . Previous studies have used changes in this score as at test of effectiveness of interventions successfully.
Progress to the Action stage for smoking cessation | Baseline, 6 and 9 months
  Will only be assessed among patients smoking at baseline (exploratory analysis; study is not powered to find significance)
Change in Well-Being | Baseline, 6 and 9 months
  Change in well-being will be computed by taking the difference in the Cantril Self-Anchoring Scale (Cantril, 1965) from baseline to 12 months follow-up. The measure asks participants to imagine a ladder with steps numbered from zero to ten, with the top representing the best possible life and the bottom representing the worst possible life, and to indicate where they feel their life falls currently and where it will be in five years.
Progress to the Action stage for drinking within recommended limits | Baseline, 6 and 9 months
  Will only be assessed among patients exceeding recommended limits at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for meeting national guidelines for physical activity | Baseline, 6 and 9 months
  Will only be assessed among patients not meeting national guidelines for physical activity at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for managing depression | Baseline, 6 and 9 months
  Will only be assessed among patients with at least mild depression (PHQ-8 score of 5 or higher) at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for drug use | Baseline, 6 and 9 months
  Will only be assessed among those indicating drug use at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage sleep management | Baseline, 6 and 9 months
  Will only be assessed among patients not meeting recommended hours at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage stress management | Baseline, 6 and 9 months
  Will only be assessed among patients not managing their stress effectively at baseline (exploratory analysis; study is not powered to find significance)
Change in level of depression | Baseline, 6 and 9 months
  Will be assessed using the Patient Health Questionnaire (PHQ-8) (Kroenke, Strine, Spritzer, Williams, Berry, & Mokdad, 2009) only among patients with at least mild depression (PHQ-8 score of 5 or higher) at baseline (exploratory analysis; study is not powered to find significance)
WHO-5 Well-being Index | Baseline, 6 and 9 months
  The 5-item World Health Organization Well-Being Index (WHO-5) is among the most widely used questionnaires assessing subjective psychological well-being.
Brief Resilience Scale (BRS) | Baseline, 6 and 9 months
  The BRS is a reliable means of assessing resilience as the ability to bounce back or recover from stress.

OTHER OUTCOMES:
Personal Financial Wellness Scale™ (PFW Scale™) | Baseline, 6 and 9 months
  The Personal Financial Wellness Scale™ (PFW Scale™) is an eight-question, self-report measure of perceived financial distress and financial well-being. The instrument measures how people are doing along a continuum extending from negative to positive feelings about and reactions to their financial situations. The tool has been scientifically determined to be a valid and reliable measure of personal financial wellness.
Mindful Attention Awareness Scale (MAAS), trait version | Baseline, 6 and 9 months
  The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place.
AUDIT-C | Baseline, 6 and 9 months
  Alcohol Use Disorders Identification Test-Consumption (AUDIT-C): a three-item scale used to assess drinking severity and as an indicator of dependence.
Personal Wellbeing Index (PWI) | Baseline, 6 and 9 months
  The PWI scale contains seven items of satisfaction, each one corresponding to a quality of life domain as: standard of living, health, achieving in life, relationships, safety, community-connectedness, and future security.
Current Tobacco Use Status | Baseline, 6 and 9 months
  Assessment of current tobacco use (all forms)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry E. Evers, PhD, Principal Investigator — Pro-Change Behavior Systems, Inc.
Locations (4):
- United States (4):
  - RallyPoint.com, Watertown, Massachusetts
  - Military Media Inc., Poughkeepsie, New York
  - Pro-Change Behavior Systems, Inc., South Kingstown, Rhode Island
  - Pilot Media, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] Humeniuk R, Ali R, Babor TF, Farrell M, Formigoni ML, Jittiwutikarn J, de Lacerda RB, Ling W, Marsden J, Monteiro M, Nhiwatiwa S, Pal H, Poznyak V, Simon S. Validation of the Alcohol, Smoking And Substance Involvement Screening Test (ASSIST). Addiction. 2008 Jun;103(6):1039-47. doi: 10.1111/j.1360-0443.2007.02114.x. Epub 2008 Mar 28. PMID 18373724
- [Background] Humeniuk, R., Dennington, v., ali R., The Effectiveness of a brief Intervention for Illicit Drugs Linked to the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) in Primary Health Care Settings: A Technical Report of Phase III Findings of the WHO ASSIST Randomized Controlled Trial. Geneva: World Health Organization. 2008. Available at http://www.who.int/substance_abuse/activities/assist_techhnicalreport_phase3_final.pdf (access 24 February 2015).
- [Background] Evers KE, Prochaska JO, Johnson JL, Mauriello LM, Padula JA, Prochaska JM. A randomized clinical trial of a population- and transtheoretical model-based stress-management intervention. Health Psychol. 2006 Jul;25(4):521-9. doi: 10.1037/0278-6133.25.4.521. PMID 16846327
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Prochaska JO, DiClemente CC, Velicer WF, Rossi JS. Standardized, individualized, interactive, and personalized self-help programs for smoking cessation. Health Psychol. 1993 Sep;12(5):399-405. doi: 10.1037//0278-6133.12.5.399. PMID 8223364
- [Background] Prochaska J, Prochaska J, Prochaska J. Building a science for multiple-risk behavior change. In: Riekert KA, Ockene JK, Pbert L, editors. The handbook of health behavior change. 4 ed. New York: Springer; 2014. p. 245-67.
- [Background] Prochaska JO, Redding C, Evers K. The Transtheoretical model and stages of change. In: Glanz K, Rimer BK, Viswanath K, editors. Health Behavior and Health Education: Theory, Research and Practice. 4 ed. San Francisco, CA: Jossey-Bass; 2008. p. 97-122.